CLINICAL TRIAL: NCT05359055
Title: An Open-label, Fixed Sequence Study to Evaluate the Effects of Multi-dose of Itraconazole or Rifampin on the Pharmacokinetic Profiles of Single Dose of SPH3127 in Healthy Volunteers
Brief Title: Drug-drug Interaction Study of SPH3127
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Shanghai Pharmaceuticals Holding Co., Ltd (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SPH3127-104
Record Dates: First submitted 2022-04-27; First posted 2022-05-03 (Actual); Last update posted 2022-07-29 (Actual); Status verified 2022-07

CONDITIONS: Drug Drug Interaction
MeSH Terms: interventions — SPH3127; Itraconazole; Rifampin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cohort 1 (Experimental): SPH3127 tablet, Itraconazole
  Interventions: Drug: SPH3127 tablet; Drug: Itraconazole
- Cohort 2 (Experimental): SPH3127 tablet, Rifampin
  Interventions: Drug: SPH3127 tablet; Drug: Rifampin

INTERVENTIONS:
Drug: SPH3127 tablet — 100mg once daily on Day 1 and Day 8
  Arms: Cohort 1
Drug: Itraconazole — 200mg once daily from Day 3 to Day10.
  Arms: Cohort 1
Drug: SPH3127 tablet — 200mg once daily on Day 1 and Day 12.
  Arms: Cohort 2
Drug: Rifampin — 600mg once daily from Day 3 to Day13.
  Arms: Cohort 2

SUMMARY:
A single center, open-label, fixed sequence Phase 1, drug-drug interaction (DDI) study in male healthy subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Willing and able to provide written informed consent;
2. Chinese Male ≥18 and ≤45 years；
3. BMI≥18.5 and ≤26.0 kg/m2 and a weight ≥50.0 kg;
4. Normal or no clinically significant diseases captured in the medical history or evidence of clinically significant findings on the vital signs, physical examination, clinical laboratory tests, and 12-lead ECG.
5. Subjects agreed to have no family planning during the study period and within 6 months after the last study drug administration, voluntarily take effective contraceptive measures and have no sperm donation plan. Non-drug contraceptive measures will be used voluntarily during the trial.
6. Subjects can communicate well with investigators, understand and comply with the requirements of this trial.

Exclusion Criteria:

1. Patients with diseases that need to be excluded, not limited to diseases of the nervous system, cardiovascular system, blood and lymphatic system, immune system, kidney, liver, gastrointestinal system, respiratory system, metabolism, bone, and other systems;
2. History of allergic diseases;
3. History of dysphagia or any gastrointestinal illness that affects drug absorption;
4. Participated in clinical trials of other investigational drugs within 3 months prior to initial administration of the investigational drug;
5. People who drink excessive tea, coffee and/or caffeinated beverages every day within 3 months before screening;
6. Prescribed medications, over-the-counter medications, dietary supplements, or Chinese herbal medicines were taken within 14 days prior to initial administration of the study drug;
7. Unwilling to avoid vigorous exercise from 48 hours before the first administration of the study drug to the end of the study;
8. Used of any drug that inhibits or induces hepatic metabolism of the drug in the 28 days prior to taking the study drug.
9. Those who have special dietary requirements and cannot follow a uniform diet;
10. Assessed by the investigators as unsuitable for participating in the study.

Ages: 18 Years to 45 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2021-12-13 (Actual); Primary Completion 2022-01-21 (Actual); Study Completion 2022-01-21 (Actual)

PRIMARY OUTCOMES:
Maximum serum concentration (Cmax) of SPH3127 | Up to 14 days
  To characterize the PK (Pharmacokinetics) of SPH3127
Area under the serum concentration-time curve (AUC) of the Dosing Interval (0-Last) of SPH3127 | Up to 14 days
  To characterize the PK (Pharmacokinetics) of SPH3127
Area under the serum concentration-time curve (AUC) of the Dosing Interval (0-infinity) of SPH3127 | Up to 14 days
  To characterize the PK (Pharmacokinetics) of SPH3127

SECONDARY OUTCOMES:
Number of subjects with adverse event. | Up to 42 days
  Adverse events, 12-lead ECG, clinical laboratory tests, physical examination and vital signs.
Time of maximum serum concentration (Tmax) SPH3127 | Up to 14 days
  To characterize the PK (Pharmacokinetics) of SPH3127
Half-life (t1/2) of SPH3127 | Up to 14 days
  To characterize the PK (Pharmacokinetics) of SPH3127
Apparent oral clearance (CL/F) of SPH3127 | Up to 14 days
  To characterize the PK (Pharmacokinetics) of SPH3127
Apparent oral volume of distribution (Vz/F) of SPH3127 | Up to 14 days
  To characterize the PK (Pharmacokinetics) of SPH3127

CONTACTS AND LOCATIONS:
Overall Officials: Qin Yu, Principal Investigator — West China Second University Hospital
Locations (1):
- West China Second University Hospital, Sichuan University, Chengdu, Sichuan, China